CLINICAL TRIAL: NCT04610710
Title: Comparing Impact of Operation and Fertility Treatment on Fertility for Women with Deep Infiltrating Endometriosis: a Multicenter Randomized Controlled Trial
Brief Title: Impact of Operation on Fertility for Women with Severe Endometriosis
Acronym: EFFORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Horsens Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Clinique Tivoli Ducos (Other)
Responsible Party: Principal Investigator, Ulla Breth Knudsen, Professor, Horsens Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Horsens MR
Record Dates: First submitted 2020-10-22; First posted 2020-10-30 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Deep Endometriosis; Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trail (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Operation (Active Comparator): Operation for severe endometriosis
  Interventions: Procedure: Operation
- Fertility treatment (Active Comparator): Fertility treatment for women with severe endometriosis.
  Interventions: Procedure: Fertility treatment

INTERVENTIONS:
Procedure: Operation — Operation for deep infiltrating endometriosis
  Arms: Operation
Procedure: Fertility treatment — In vitro fertilisation (IVF) and IVF-intracytoplasmic injection (ICSI)
  Arms: Fertility treatment

SUMMARY:
The EFFORT study compares the impact on fertility of operation or fertility treatment (IVF, in vitro fertilization) in a multicenter randomized controlled trial. The study population consists of women with colorectal deep infiltrating endometriosis and a pregnancy intention. These women will be randomized to either of the two treatment groups: Group A = Operation or Group B = fertility treatment (IVF). Group A will be further divided postoperatively into spontaneous conception or IVF depending on the Endometriosis Fertility Index score.

ELIGIBILITY:
Inclusion Criteria:

* Rectosigmoid endometriosis and wish for surgery
* Pregnancy intention for at least 6 months
* AMH above 5 pmol/ml
* Maximum of 2 previous IVF treatments
* Male partner

Exclusion Criteria:

* Endometriosis involving the ureter unilaterally or bilaterally (randomization unethical)
* BMI above 32
* Contraindication for IVF (untreated uterine factor infertility, untreated/maltreated systemic or malignant disease, oocyte aspiration severely riskful (e.g. severe abdominal adhesions)
* No wish for randomization

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 352 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2035-07-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative pregnancy rate (CPR) | 18 months
  Rate of cumulative pregnancies defined as a fetal heartbeat by ultrasound at gestational week 6 to 8
Live birth rate (LBR) | 18 months
  Rate of live births

SECONDARY OUTCOMES:
Non-viable pregnancies | 18 months
  Number of biochemical pregnancies, miscarriages, missed abortions, extrauterine pregnancies and pregnancies of unknown location (PUL)
Ovarian potential | Baseline and 9-18 months
  Concentration of Anti-Müllerian hormone (AMH)
Time to pregnancy | 18 months
  Shortest time from intervention date to date of visualisation of the first ongoing pregnancy
Postoperative complications | 18 months
  Rate of complications in accordance to Clavien-Dindo Classification, including anastomotic leakage or stenosis, ureteral lesion or obstruction, pelvic abscess, fistula, bladder or bowel perforation and urinary retention
Fertility treatment complications | 18 months
  Rate of hospital admissions, bleeding, superinfection, worsening of pain or having ovarian hyperstimulation syndrome (OHSS)
Pain score | Baseline, 9 and 18 months
  Numeric Rating Scale (NRS) score from 0 to 10, where 10 implies the worst pain
Quality of Life (QoL) | Baseline, 9 and 18 months
  Development in Endometriosis Health Profile (EHP-30+23), including section C (sexual function QoL questions) and section F (fertility QoL questions)
Delayed bowel function | Baseline, 9 and 18 months
  Development in bowel function rated by Low Anterior Resection Syndrome (LARS) score
Delayed bladder function | Baseline, 9 and 18 months
  Development in urinary tract function rated by International Consultation on Incontinence Questionnaire (ICIQ- FLUTS)
Endometriosis hormonal and inflammatory status | Baseline and 9-18 months
  Concentrations of hormonal and inflammatory markers in blood samples
Follicles, oocytes, fertilized oocytes, blastocysts, and frozen embryos | 18 months
  Number of follicles as measured at last scan prior to oocyte pick-up (OPU), number of oocytes at OPU, fertilized oocytes, blastocysts and frozen embryos
Blastocyst morphology score | 18 months
  Gardner scoring system, Steer grading system, Veecks criteria, or other scoring systems of blastocyst morphology

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N, Central Region
  - Horsens Regional Hospital, Horsens, Central Region
- The Endometriosis Center, Clinique Tivoli-Ducos, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raos M, Roman H, Seyer-Hansen M, Kesmodel US, Knudsen UB. EFFORT study: Comparing impact of operation and assisted reproductive technologies on fertility for women with deep infiltrating endometriosis - study protocol for a multicentre randomised trial. BMJ Open. 2022 Apr 11;12(4):e052877. doi: 10.1136/bmjopen-2021-052877. PMID 35410921